CLINICAL TRIAL: NCT01850368
Title: Multicenter Phase II Study of Stereotactic Ablative Radiotherapy for Hepatocellular Carcinoma With Major Portal Vein Invasion
Brief Title: Stereotactic Ablative Radiotherapy for Hepatocellular Carcinoma With Major Portal Vein Invasion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Cancer Center Hospital (Other)
Collaborators: Seoul National University Hospital (Other); Dongnam Institute of Radiological & Medical Sciences (Other); Soon Chun Hyang University (Other); Inha University Hospital (Other); Incheon St.Mary's Hospital (Other); Gyeongsang National University Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Mi-Sook Kim, Doctor, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-1209-001-007; KCT0000542 (Registry Identifier: Clinical Research Information Service); KROG 13-02 (Registry Identifier: Korean Radiation Ocology Group); K-1209-001-007 (Other: Korea Institute of Radiological & Medical Science IRB)
Record Dates: First submitted 2013-05-02; First posted 2013-05-09 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombus
Keywords: Hepatocellular carcinoma; Stereotactic ablative radiotherapy; Stereotactic body radiotherapy; Portal vein tumor thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic ablative radiotherapy (Experimental): Stereotactic ablative radiotherapy for HCC patients with major portal vein tumor thrombosis (tumor thrombosis in the main portal vein or 1st branch of portal vein)
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — The HCC patients with major portal vein tumor thrombosis (tumor thrombosis in the main portal vein or 1st branch of portal vein) will be included in this study. Total stereotactic ablative radiotherapy (SABR) doses will be 40 Gy in 4 fractionations. Patients receive 4 fractionations separated by >48 hours.
  At least 700 ml of normal liver (entire liver minus cumulative GTV) should not receive a total dose of > 19.2 Gy in three fractions. If volume of normal liver does not exceed 700 ml, at least 70% of normal liver should not receive a total dose of > 19.2 Gy. Dose of spinal cord do not exceed 26 Gy. Dose of esophagus, stomach and intestine do not exceed 35 Gy.
  Other Names: Stereotactic body radiotherapy

SUMMARY:
Recently, several studies reported promising outcomes of patients after external beam radiotherapy (EBRT) for hepatocellular carcinoma (HCC) with portal vein tumor thrombosis. However, conventional EBRT is composed of many fractions (20-35 fractions). On the other hand, stereotactic ablative radiotherapy is a newly emerging treatment method to deliver a high dose of radiation to the target using a few fractions with a high precision within body. SABR increases radiation biologic effect for tumor, makes patients more comfortable due to reduction of the number of hospital visit, and enables patients to receive another treatment more quickly. This study will evaluate SABR effect with 40 Gy in 4 fractions for HCC with major portal vein tumor thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 20 years of age
* Initially diagnosed or recurrent hepatocellular carcinoma (HCC)
* Eastern Cooperative Oncology Group performance status 0 or 1
* HCC with major portal vein tumor thrombosis (tumor thrombosis in the main portal vein or 1st branch of portal vein)
* Cirrhotic status of Child Pugh class A or B7
* Patients can have extra-hepatic disease; provided the hepatic disease is the highest burden, the extra-hepatic disease is low burden and potentially treatable with radiotherapy, chemotherapy and target agent etc; patient survival is expected to be at least 6 months.
* Patient or guardian must be able to provide verbal and written informed consent

Exclusion Criteria:

* Prior trans-arterial chemo-embolization ≥4 after diagnosis of major portal vein tumor thrombosis
* Severe complication caused by liver cirrhosis eg. variceal bleeding, poorly controlled ascites, hepatic encephalopathy)
* Uncontrolled inter-current illness except liver cirrhosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Tumor stabilization rate | 2 months
  Tumor stabilization rate was based on the combined number of patients with complete response(CR), partial response(PR), and stable disease(SD) by modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.

SECONDARY OUTCOMES:
Overall survival | 6 months, 1 year and 2 year
  From the date of SABR to the date of death or last follow-up
Tumor progression free survival | 6 months, 1 year and 2 year
  From the date of SABR to the date of first failure or last follow-up
Treatment related toxicity | 1 year
  Adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0; Classic radiation induced liver disease; Non-classic Classic radiation induced liver disease; Worsening of Child-Turcotte-Pugh score; Worsening of MELD score

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Sook Kim, MD, PhD, Principal Investigator — Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences
Locations (8):
- South Korea (8):
  - Gyeongsang National University Hospital, Jinju, Gyeongsang-nam-do
  - Dongnam Institute of Radiological & Medical Sciences, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Catholic University Incheon St. Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoon SM, Lim YS, Won HJ, Kim JH, Kim KM, Lee HC, Chung YH, Lee YS, Lee SG, Park JH, Suh DJ. Radiotherapy plus transarterial chemoembolization for hepatocellular carcinoma invading the portal vein: long-term patient outcomes. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):2004-11. doi: 10.1016/j.ijrobp.2011.03.019. Epub 2011 May 27. PMID 21621346
- [Background] Kim JY, Chung SM, Choi BO, Kay CS. Hepatocellular carcinoma with portal vein tumor thrombosis: Improved treatment outcomes with external beam radiation therapy. Hepatol Res. 2011 Sep;41(9):813-24. doi: 10.1111/j.1872-034X.2011.00826.x. Epub 2011 Jun 22. PMID 21696524
- [Background] Tanaka A, Morimoto T, Yamaoka Y. Implications of surgical treatment for advanced hepatocellular carcinoma with tumor thrombi in the portal vein. Hepatogastroenterology. 1996 May-Jun;43(9):637-43. PMID 8799408
- [Background] Kang JK, Kim MS, Cho CK, Yang KM, Yoo HJ, Kim JH, Bae SH, Jung DH, Kim KB, Lee DH, Han CJ, Kim J, Park SC, Kim YH. Stereotactic body radiation therapy for inoperable hepatocellular carcinoma as a local salvage treatment after incomplete transarterial chemoembolization. Cancer. 2012 Nov 1;118(21):5424-31. doi: 10.1002/cncr.27533. Epub 2012 May 8. PMID 22570179
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977